CLINICAL TRIAL: NCT05974813
Title: The Effect of Short-term L-citrulline Supplementation on Blood Pressure and Arterial Stiffness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: European University Cyprus (Other)
Responsible Party: Principal Investigator, Dr. Anastasios Theodorou, Associate Professor, European University Cyprus
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: EUC_cit
Record Dates: First submitted 2023-07-18; First posted 2023-08-03 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-07

CONDITIONS: Blood Pressure
MeSH Terms: interventions — Citrulline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- L-Citrulline (Experimental): Participants will receive 6 g (3 g every 12 h) of L-citrulline (Now, L-citrulline Pure Powder) for six-days.
  Interventions: Dietary Supplement: L-Citrulline
- Placebo (Placebo Comparator): Participants will receive 6 g (3 g every 12 h) of maltodextrin (Now, Maltodextrin) for six-days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: L-Citrulline — 6 g (3 g every 12 h) of L-citrulline for six days
  Arms: L-Citrulline
Dietary Supplement: Placebo — 6 g (3 g every 12 h) of maltodextrin for six days
  Arms: Placebo

SUMMARY:
The goal of this clinical trial is to examine the effect of short-term L-Citrulline on central and peripheral blood pressure in healthy older adults. The main questions it aims to answer are:

* Does L-citrulline favorably affect blood pressure at rest and during exercise?
* Does L-citrulline favorably affect arterial stiffness?
* Does L-citrulline favorably affect muscle oxygenation at rest and during exercise?

Participants will be asked to consume L-citrulline and a placebo for six days and participate in the evaluation of their blood pressure, arterial stiffness, and muscle oxygenation before and after each intervention.

Researchers will compare L-citrulline and placebo groups to examine whether L-citrulline supplementation affects the above health parameters.

ELIGIBILITY:
Inclusion Criteria:

* subject provides written informed consent.
* normal health profile.

Exclusion Criteria:

* history of musculoskeletal injury in the legs during the previous six months.
* smoker.
* consumption of any medication the last three months.
* consumption of any nutritional supplement the last three months.

Ages: 55 Years to 70 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 12 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Change in aortic and brachial systolic blood pressure (rest) | Change from baseline aortic and brachial systolic blood pressure at 7 days.
Change in aortic and brachial systolic blood pressure | Change from baseline aortic and brachial systolic blood pressure at the second minute of exercise.
Change in carotid-femoral pulse wave velocity (cfPWV) (rest) | Change from baseline aortic and brachial systolic blood pressure at 7 days.

SECONDARY OUTCOMES:
Change in pulse pressure (rest) | Change from baseline pulse pressure at 7 days.
Change in heart rate (rest) | Change from baseline heart rate at 7 days.
Change in augmented pressure (rest) | Change from baseline augmented pressure at 7 days.
Change in augmentation index (rest) | Change from baseline augmentation index at 7 days.
Change in forward and backward wave pressure (rest) | Change from baseline forward and backward wave pressure at 7 days.
Change in muscle oxyhemoglobin (rest) | Change from baseline oxyhemoglobin at 7 days.
Change in pulse pressure (exercise) | Change from baseline pulse pressure at the second minute of exercise.
Change in heart rate (exercise) | Change from baseline heart rate at the second minute of exercise.
Change in augmented pressure (exercise) | Change from baseline augmented pressure at the second minute of exercise.
Change in augmentation index (exercise) | Change from baseline augmentation index at the second minute of exercise.
  The ideal augmentation index is between 20 and 80. Values above 80 are considered high, and above 121 indicate high arterial stiffness.
Change in forward and backward wave pressure (exercise) | Change from baseline forward and backward wave pressure at the second minute of exercise.
Change in muscle deoxyhemoglobin (exercise) | Change from baseline muscle deoxyhemoglobin at the second minute of exercise.
Change in muscle deoxyhemoglobin (rest) | Change from baseline muscle deoxyhemoglobin at 7 days.
Change in muscle oxyhemoglobin (exercise) | Change from baseline muscle oxyhemoglobin at the second minute of exercise.
Change in muscle oxyhemoglobin (rest) | Change from baseline muscle oxyhemoglobin at 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Marios Vryonides, Dr., Study Director — European University Cyprus
Locations (1):
- European University Cyprus, Nicosia, Cyprus

IPD SHARING:
Plan to Share IPD: No